CLINICAL TRIAL: NCT06154889
Title: Rehabilitation by Multifactorial Approach After a Latarjet Procedure : Prospective Single-center Randomized Study (MATASI-L)
Brief Title: Rehabilitation by Multifactorial Approach After a Latarjet Procedure
Acronym: MATASI-L
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Générale dAnnecy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A02057-38
Record Dates: First submitted 2023-11-21; First posted 2023-12-04 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Dislocation Shoulder
Keywords: shoulder instability; kinesiophobia; Latarjet; apprehension
MeSH Terms: conditions — Shoulder Dislocation; Kinesiophobia | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Convention readaptation protocol (Active Comparator): Patients have a conventional re-education after surgery for anterior shoulder dislocation (Latarjet procedure)
  Interventions: Other: Conventional reeducation
- Readaptation protocol with psychologic intervention (Experimental): Patient have a conventional re-education after surgery for anterior shoulder dislocation (Latarjet procedure) with addition of 4 consultations with a sports psychologist
  Interventions: Other: consultations with a psychologist

INTERVENTIONS:
Other: consultations with a psychologist — Consultations with a sports psychologist to decrease kinesiophobia
  Arms: Readaptation protocol with psychologic intervention
Other: Conventional reeducation — Conventional reeducation
  Arms: Convention readaptation protocol

SUMMARY:
Kinesiophobia (fear of physical movement) is common after a previous shoulder dislocation and persists after one year, regardless of the occurrence of a recurrence. This kinesiophobia is associated with a lower level of physical activity and a lower return to sport. Increased kinesiophobia, combined with other psychological factors such as depression and fear of re-injury in patients with shoulder instability, results in poor outcomes after treatment. Given that there is currently no postoperative protocol that takes this psychological component into account, a new rehabilitation protocol focused on reducing kinesiophobia was recently designed as part of an international consensus study based on the method Delphi. This protocol includes a core set of evidence-based interventions aimed at regaining functional stability of the shoulder and reducing fear of recurrent dislocation and kinesiophobia. The goal of this study is to determine if we can reduce kinesiophobia in patients who have undergone stabilization surgery for anterior shoulder instability using this new rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Primary or recurrent traumatic anterior dislocation of the shoulder
2. Indication of abutment according to Latarjet (arthroscopic or open sky)
3. Age: 18-67 years
4. Understanding of the French language spoken and written
5. Written informed consent (in accordance with to ICH-GCP guidelines)

Exclusion Criteria:

1. Posterior or multidirectional instability of the shoulder (Beighton score >5)
2. Age <18 or >67 years.
3. Patients with additional rotator cuff tear.
4. Patients with a history of surgery on either shoulder.
5. Patients with connective tissue disorders (eg Ehler-Danlos).
6. Patients with (current) anxiety disorders or using anxiolytic medications (eg, antipsychotics) (criterion based on patient record/indications).
7. Patients with neurological disorders or systemic disease.
8. Patients with inflammatory disease, rheumatoid arthritis or active malignancy.
9. Patients previously hospitalized for shoulder pain
10. Patients with upper tubercle fracture
11. Patients with motor neurological deficit
12. Pregnant or breastfeeding patient
13. Patient protected under protective measure

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability Index (WOSI) | 6 months
  self-evaluating shoulder instability quality of life score : 21 items. The patient is asked to grade the function of a specific item on a horizontal visual analog scale from 0 to 100 mm.
  Each question results in a number between 0 and 100 and the total score may be presented as a number between 0 and 2,100 points (where 0 represents no deficit and 2,100 the worst)

SECONDARY OUTCOMES:
Shoulder subjective value | 6 months
  subjective evaluation by the patient of shoulder function, expressed as a percentage of a normal shoulder. This score ranges from 0 to 100%.
ability to return to work | 6 months
  time indication
ability to return to sport | 6 months
  time indication
Patient's pain | 6 months
  visual analogic scale between 0 and 10
Patient's kinesiophobia | 6 months
  Tampa's scale : 17 questions with scored results between 1 and 4
S-starts test (including psychologic evaluation) | 6 months
  Composite score :
  * Shoulder Instability-Return to Sport after Injury questionnaire (12 items each assessed on a scale from 0 to 10) quantifying the psychological readiness of athletes to return to sport following shoulder instability through evaluating emotions, confidence in performance, and perceived risk
  * 4 physical performance tests
  * Maximal Isometric Strength of Glenohumeral Rotator Muscles
  * Y Balance Test for Upper Extremity
  * Modified Closed Kinetic Chain Upper Extremity Stability Test
  * Unilateral Seated Shot Put Test

CONTACTS AND LOCATIONS:
Overall Officials: Geert Alexander Buijze, MD, Principal Investigator — Clinique Générale d'Annecy
Locations (1):
- Clinique Générale d'Annecy, Annecy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soares MN, Shirinskiy IJ, Schachner J, Matasi Collaborator Group MCG, Macken AA, Kling A, Lafosse T, van den Bekerom MPJ, Buijze GA. Multifactorial approach training for anterior shoulder instability after a Latarjet procedure: protocol for a randomised controlled trial. BMJ Open. 2026 Jan 21;16(1):e109378. doi: 10.1136/bmjopen-2025-109378. PMID 41565337